CLINICAL TRIAL: NCT06030362
Title: Double Blinded Placebo Controlled Feasibility Study to Evaluate a Combination Probiotic in Adults With Obesity
Brief Title: Probiotic Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arpana Church, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 22-000796
Record Dates: First submitted 2023-08-04; First posted 2023-09-11 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Food Addiction
Keywords: Probiotic; Dietary Supplement
MeSH Terms: conditions — Obesity; Food Addiction | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dietary Supplement taken once daily for 3 months (90 days).
  Arms: Probiotic
Dietary Supplement: Placebo — Dietary Supplement taken once daily for 3 months (90days).
  Arms: Placebo

SUMMARY:
The current standard of care for obesity is the optimal management of comorbid conditions such as diabetes and hyperlipidemia, and counseling on diet, weight loss, or increased physical activity programs. However, lifestyle, diet, and behavioral interventions may provide between 7-10% reduction in initial weight and even fewer with long-term weight loss. In severely obese patients (BMI>40 or BMI>35 with comorbidities), bariatric surgery is also a potential treatment, but there is a high barrier for patients to undergo surgery for weight loss. These barriers include an aversion to major abdominal surgery, long recovery time, potential risk of vitamin deficiency, and risk for abdominal pain. For these reasons, there is a paramount need for other treatments for obesity and for food addiction.

The current standard of care for obesity and food addiction is difficult to implement and lacks sustained efficacy. Most struggle to complete treatment, lose minimal weight, lack sustained weight loss, and engage in the well-known "YoYo" diet phenomenon. While bariatric surgery is currently the only effective treatment for obesity, there are several barriers associated with it such as eligibility requirements, invasiveness, difficult recovery, and cost making it not readily available for everyone. Some approved medications that help with obesity, such as orlistat, lorcaserin, or naltrexone-bupropion, have not been widely adopted by providers or patients due to their limited responses and adverse side effects. Probiotic cocktails have shown to be safe with little to no side effects. Preclinical models of probiotics demonstrate the ability to curb obesity in animal models. Therefore, a probiotic that is able to show significant weight loss along with lifestyle modifications would be highly adopted and desirable.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* BMI 25-40
* Male and Female
* Not Pregnant or Nursing

Exclusion Criteria:

* Co-morbidities including but not limited to:
* Type 1 (insulin dependent) diabetes
* vascular disease
* drastic weight loss (more than 10lbs over the preceding 2months)
* frequent strenuous exercise (i.e. marathon runners/heavy weight lifting)
* abdominal surgeries including weight loss surgery or partial/complete resection of stomach or bowel
* untreated thyroid disease
* neurological disease
* Major medical condition the PI/MD feels would put the subject at risk or interfere with data collection.
* Chronic pain
* Diagnosed DSM IV active psychiatric illness including eating disorders. Must not be active or present for at least 2 years. Participants with a positive endorsement on the MINI+ will be excluded.
* Using medications known to affect hunger/satiety/appetite
* Pregnant, lactating, postpartum less than 6months.
* Women of childbearing potential who are not practicing birth control or are planning to get pregnant during the study.
* Use of oral/IV antibiotics within the last 3 months
* Use of probiotics in the last 3 months.
* Heavy use of alcohol and drugs will be determined by a positive endorsement on the MINI+. If the MINI+ is positive for alcohol or drug dependence or abuse, the participant will be excluded. In regards to tobacco use, participants will be excluded if they smoke more than 1/2 pack per day.
* Cannabis use will not be exclusionary. If the MINI+ is positive for drug dependence or abuse, the participant will be excluded.
* Significant change in usual diet and/or weight loss of more than 10lbs in the last 2 months.
* Anyone taking medicines on the medication exclusion list.
* Non-English Speakers (due to the use of validated questionnaires and limited availability of translated copies, participants must be fluent in English so that they will be able to read and follow directions easily.
* Maintenance pharmacotherapies will not be exclusionary so long as they have been on a stable dose for 6months.
* Body weight at enrollment greater than 400lbs.
* Exclude from Optional MRI if: participant is unable to safely participate in the MRI (claustrophobia, presence of devices affected by MRI such as pacemakers, neurostimulators, metallic foreign bodies, etc.).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences in metabolite concentrations pre & post intervention - Stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (week 6), and once at the final 3month appointment (week 12).
  Measurement of metabolomics via stool specimen.
Differences in metabolite concentrations pre & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (week 6), and once at the final 3month appointment (week 12).
  Measurement of metabolomics via blood specimen.
Differences in microbiome levels pre & post intervention - Stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (week 6), and once at the final 3month appointment (week 12).
  16S RNA sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (week 6), and once at the final 3month appointment (week 12).
  16S RNA sequencing to measure microbiome levels via blood specimen.
Differences in microbiome levels pre & post intervention - Stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (week 6), and once at the final 3month appointment (week 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (week 6), and once at the final 3month appointment (week 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via blood specimen.

SECONDARY OUTCOMES:
Differences in Subjective Stress Response - PANAS | Lasting approximately 10 minutes, measured pre & post the laboratory stress tasks, at baseline (week 0) and end of study (week 12).
  Between and within group differences on the negative affect subscale from the Brief Positive Affect and Negative Affect Scale (PANAS) before and after the laboratory stress tasks. PANAS scores can range from 10-50 for both the positive and negative affect, with the lower scores representing lower levels of positive/negative affect, and higher scores representing higher levels of positive/negative affect.
Changes in Autonomic Measures - Heart Rate Variability | Measured throughout each laboratory stress task during the baseline (week 0) and end of study (week 12) visits, lasting approximately 1 hour.
  Between and within group differences in overall average change in heart rate variability pre and post each laboratory stress task.
Changes in Autonomic Measures - Skin Conductance | Measured throughout each laboratory stress task during the baseline (week 0) and end of study (week 12) visit. Lasting approximately 1 hour.
  Between and within group differences in overall average change in skin conductance response (SCR) pre and post each laboratory stress task measured using BIOPAC GSR (galvanized skin response) 100C system. Measured in Hz.
Changes in Autonomic Measures - Diastolic & Systolic blood pressure | Measured throughout each laboratory stress task during the baseline (week 0) and end of study (week 12) visit. Lasting approximately 1 hour.
  Between and within group differences in overall average change in both diastolic and systolic blood pressure pre and post each laboratory stress task.
Differences in Attention/Executive Function - Color Stroop | Lasting approximately 10minutes, measured at baseline (week 0) and end of study (week 12).
  Between and within group differences on the time it takes to complete the Color Stroop attention/executive function lab stress task.
Differences in Attention/Executive Function - Trails A & B | Lasting approximately 10minutes, measured at baseline (week 0) and end of study (week 12).
  Between and within group differences on the time it takes to complete the Trails A & B attention/executive function lab stress task.
Differences in Emotional Arousal System - IAPS task | Lasting approximately 15minutes, measured at baseline (week 0) and end of study (week 12).
  Between and within group differences in valence and emotional arousal ratings during the International Affective Picture System (IAPS) task.
Systolic and Diastolic Blood Pressure | Measured three times, once at each in-clinic appointment (week 0, week 6, week 12).
  Measurement of the pressure of circulating blood at rest
Anthropometrics - BMI | Measured three times, once at each in-clinic appointment (week 0, week 6, & week 12)
  Measurement of height(in) & weight(lbs), used to calculate body mass index (BMI).
Questionnaire Data - Diet | Self-Reported by the participant at home, collected 3 times (1) before beginning the dietary supplement, (2) at least 1 week before the mid-study appointment, and (3) within 1 week of finishing the 90-day dietary supplement.
  Use of validated surveys including the Food Frequency questionnaire, Food Choice Questionnaire.
Questionnaire Data | Self-Reported by the participant at home, collected 3 times (1) before beginning the dietary supplement, (2) at least 1 week before the mid-study appointment, and (3) within 1 week of finishing the 90-day dietary supplement.
  Use of validated surveys to assess ingestive behaviors, stress, health, physical activity, etc.
Anthropometrics - waist and hip circumference | Measured three times, once at each in-clinic appointment (week 0, week 6, & week 12)
  Measurement of waist and hip circumference (cm).

OTHER OUTCOMES:
Differences in Multimodal Brain Signatures | Optional - Measured twice, once at baseline (week 0) and once at end of study (week 12) visit. Lasting approximately 1.5hours.
  Neuroimaging of a subset of participants brain via magnetic resonance imaging (MRI) procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Arpana Gupta, PhD, Principal Investigator — The Regents of the University of California, Los Angeles; Tien Dong, MD, PhD, Principal Investigator — The Regents of the University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to make the de-identified data available for sharing with other researchers.